CLINICAL TRIAL: NCT02053181
Title: A Phase 1, Open-label, Single Oral Dose Study to Investigate the Pharmacokinetics, Safety, and Tolerability of Cadazolid in Patients With Severe Clostridium Difficile Infection (CDI)
Brief Title: Study to Investigate the Pharmacokinetics and Safety of Cadazolid in Patients With Clostridium Difficile Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: AC-061-103
Record Dates: First submitted 2014-01-30; First posted 2014-02-03 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Clostridium Difficile Infection
Keywords: Cadazolid; ACT-179811; Pharmacokinetics; Safety; Tolerability
MeSH Terms: conditions — Clostridium Infections | interventions — cadazolid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cadazolid (Experimental): Single oral dose of 3000 mg.
  Interventions: Drug: Cadazolid

INTERVENTIONS:
Drug: Cadazolid — Cadazolid was provided as dry powder for oral suspension (Amber glass bottles of 60 mL). The powder was reconstituted with tap water by a pharmacist immediately prior to dispensing to subjects.
  Other Names: ACT-179811

SUMMARY:
The study investigated the pharmacokinetics, safety, and tolerability of cadazolid in subjects with severe Clostridium difficile diarrhea (CDAD) and whether this influenced the quantity of cadazolid absorbed into the systemic circulation.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any study-mandated procedure.
* Non-pregnant females were to remain non-pregnant for 1 month after the end of the study. Female subjects of child-bearing potential must have had a negative serum pregnancy test at screening and must have used a reliable method of contraception
* Subjects with severe CDAD; Clostridium difficile infection (CDI) must have been microbiologically proven, using a validated enzyme-linked immunosorbent assay (ELISA) for the detection of C. difficile toxin A (TcdA) and/or C. difficile toxin B (TcdB). The severity of CDAD was assessed according to the current European Union guidelines - European Society of Clinical Microbiology and Infectious Diseases (ESCMID).
* Received oral vancomycin or oral/intravenous (i.v.) metronidazole therapy for the treatment of CDAD.
* Ability to communicate well with the investigator in the local language, and to understand and comply with the requirements of the study.

Exclusion Criteria:

* Known hypersensitivity to any excipients of the drug formulation.
* Clinical evidence of any relevant disease other than CDAD and/or existence of any surgical or medical condition that might interfere with the absorption, distribution, metabolism or excretion of the study drug.
* Veins unsuitable for i.v. puncture on either arm (e.g., veins that are difficult to locate, access, or puncture; veins with a tendency to rupture during or after puncture).
* Subjects with rare hereditary fructose intolerance, glucose-galactose malabsorption, saccharase-isomaltase deficiency or previously undiagnosed diabetes mellitus.
* Subjects who have a life-threatening condition, which may be related to CDAD or other underlying illness.
* Any clinically relevant electrocardiogram (ECG) abnormality at screening.
* Subjects who were unable to swallow or have difficulty swallowing.
* Subjects with vomiting, ileus or not passing stool.
* Likelihood of death within 72 hours from any cause.
* Life-threatening or fulminant CDAD (White blood cell count > 30 × 10^9/L; temperature > 40 °C; or septic shock, peritoneal signs or significant dehydration).
* History of ulcerative colitis or Crohn's disease.
* Loss of 250 mL or more of blood within 3 months prior to screening.
* Positive results from the hepatitis serology, except for vaccinated subjects, at screening.
* Positive results from the human immunodeficiency virus (HIV) serology at screening.
* Legal incapacity or limited legal capacity at screening.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-08; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of cadazolid | 144 hours
  Blood samples for pharmacokinetic analysis taken immediately prior to dosing with cadazolid, and at 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, and 144 hours after dosing. Cmax was calculated on the basis of the blood sampling time points.
Time to reach maximum plasma concentration (tmax) of cadazolid | 144 hours
  Blood samples for pharmacokinetic analysis taken immediately prior to dosing with cadazolid, and at 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, and 144 hours after dosing. tmax was calculated on the basis of the blood sampling time points.
Area under the plasma concentration-time curve (AUC(0-144h)) of cadazolid | 144 hours
  Blood samples for pharmacokinetic analysis taken immediately prior to dosing with cadazolid, and at 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, and 144 hours after dosing. AUC(0-144) was calculated according to the linear trapezoidal rule using the measured concentration-time values above the limit of quantification.
Unchanged cadazolid in urine up to Day 7 | 144 hours
  Urine was collected into standard-weight polyethylene containers over the following time intervals: 0-12 h, 12-24 h, 24-36 h, 36-48 h, 48-72 h, 72-96 h, 96-120 h, and 120-144 h. The concentration of cadazolid was determined using validated liquid chromatography-tandem mass spectrometry assays. The amount of drug excreted in the urine was obtained by multiplying the concentration of drug by the volume of matrix collected.
Unchanged cadazolid in faeces up to Day 7 | 144 hours
  Faeces were collected in pre-weighed polypropylene boxes. The concentration of cadazolid was determined using validated liquid chromatography-tandem mass spectrometry assays. The amount of drug excreted in the faeces was obtained by multiplying the concentration of drug by the volume of matrix collected.

SECONDARY OUTCOMES:
Change from baseline up to Day 7 in systolic blood pressure (SBP) | 144 hours
  Blood pressure (systolic and diastolic) and pulse rate were measured using an automatic oscillometric device, always on the leading arm (i.e., leading arm = writing arm). Measurements were recorded in the supine position after the subject had rested for a 5-minute period.
Change from baseline up to Day 7 in diastolic blood pressure (DBP) | 144 hours
  Blood pressure (systolic and diastolic) and pulse rate were measured using an automatic oscillometric device, always on the leading arm (i.e., leading arm = writing arm). Measurements were recorded in the supine position after the subject had rested for a 5-minute period.
Change from baseline up to Day 7 in pulse rate | 144 hours
  Blood pressure (systolic and diastolic) and pulse rate were measured using an automatic oscillometric device, always on the leading arm (i.e., leading arm = writing arm). Measurements were recorded in the supine position after the subject had rested for a 5-minute period.
Change from baseline to Day 7 in body weight | 144 hours
  Body weight was measured using the same weighing scales.
Change from baseline up to Day 7 in heart rate | 144 hours
  Heart rate was determined from standard 12-lead electrocardiographs (ECGs) recorded in the supine position, after a 5-minute period of resting.
Change from baseline up to Day 7 in PQ interval (time interval from the beginning of the P wave to the beginning of the QRS complex) | 144 hours
  PQ interval was determined from standard 12-lead ECGs recorded in the supine position, after a 5-minute period of resting.
Change from baseline up to Day 7 in QRS duration (time interval from the beginning of the Q wave to the end of the S wave) | 144 hours
  QRS duration was determined from standard 12-lead ECGs recorded in the supine position, after a 5-minute period of resting.
Change from baseline up to Day 7 in QT (time interval from beginning of the Q wave until end of the T wave) | 144 hours
  QT interval was determined from standard 12-lead ECGs recorded in the supine position, after a 5-minute period of resting.
Change from baseline up to Day 7 in QT interval according to Bazett's correction (QTcB) | 144 hours
  QTcB interval was determined from standard 12-lead ECGs recorded in the supine position, after a 5-minute period of resting. The QTcB interval is the QT interval (interval from beginning of the Q wave until end of the T wave) corrected for heart rate with Bazett's formula (QTcB = QT/RR^0.5 where RR is 60/heart rate)
Change from baseline up to Day 7 in QT interval according to Fridericia's correction (QTcF) | 144 hours
  QTcF interval was determined from standard 12-lead ECGs recorded in the supine position, after a 5-minute period of resting. The QTcF interval is the QT interval (interval from beginning of the Q wave until end of the T wave) corrected for heart rate with Fridericia's formula (QTcB = QT/RR^0.33 where RR is 60/heart rate)
Frequency of treatment-emergent ECG abnormalities from up to Day 7 | 144 hours
  Treatment-emergent abnormalities were determined from standard 12-lead ECGs recorded in the supine position, after a 5-minute period of resting. An ECG abnormality was considered treatment-emergent if it was not present during the screening period and/or at time of pre-dose assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Mackie, MSc, Study Director — Actelion
Locations (1):
- Clinical Hospital for Infective Disease, Zagreb, Croatia

REFERENCES:
- [Derived] Gehin M, Desnica B, Dingemanse J. Minimal systemic and high faecal exposure to cadazolid in patients with severe Clostridium difficile infection. Int J Antimicrob Agents. 2015 Nov;46(5):576-81. doi: 10.1016/j.ijantimicag.2015.07.015. Epub 2015 Sep 3. PMID 26419191